CLINICAL TRIAL: NCT06511752
Title: Educational Support Group Program for Carepartners of Bilingual and Spanish-speaking Persons With Progressive Forms of Aphasia and for Persons With Progressive Forms of Aphasia
Brief Title: Educational Support Group Program for Bilingual and Spanish-speaking Carepartners and People With Progressive Aphasia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: The Association for Frontotemporal Degeneration (Unknown)
Responsible Party: Principal Investigator, Stephanie Grasso, Assistant Professor, University of Texas at Austin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005541
Record Dates: First submitted 2024-06-06; First posted 2024-07-22 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Dementia; Primary Progressive Aphasia; Aphasia; Progressive Aphasia; Progressive Aphasia in Alzheimer's Disease
Keywords: bilingual; Spanish; Castellano; multicultural; multilingual
MeSH Terms: conditions — Alzheimer Disease; Dementia; Aphasia, Primary Progressive; Aphasia | interventions — Self-Help Groups

STUDY DESIGN:
Intervention Model Description: Behavioral intervention- support group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Condition (Experimental): Support group meetings and strategy practice
  Interventions: Behavioral: Psychosocial educational, support group and implementation of strategies

INTERVENTIONS:
Behavioral: Psychosocial educational, support group and implementation of strategies — Psychosocial educational, support group and implementation of strategies

SUMMARY:
The current study aims to examine the benefits of an education/support group program for individuals with progressive aphasia (caused by various etiologies, diagnoses) and their carepartners. The current study utilizes pre-, post-treatment, and follow-up assessments to measure effects of a psychoeducational support group and an implementation/communication skills training phase on measures of psychosocial function, communicative effectiveness and speech/language function. Analysis of study-specific surveys and semi-structured interviews will provide qualitative data regarding outcomes. Before beginning the education and support group, focus groups will be run in order to set priorities for the themes to be included in the education program. Participants will join via tele-based means if preferred and these participants may reside in the United States, or internationally including Mexico and Spain.

DETAILED DESCRIPTION:
Two educational/support group routes will be offered:

1. Progressive aphasia (PA) educational/support group or
2. Caregiver educational support group with an implementation phase (including their partner with PA).

The caregiver educational support group path will be delivered in two phases, whereas the PA educational support group path will only consist of the first phase. The first phase of the caregiver educational support group will focus on the educational support group and the second phase will consist of implementation and practice of strategies with feedback provided by the clinician.

The educational/support groups (Routes 1 and 2) will include opportunities for discussion of issues related to language-led dementia or progressive aphasia (e.g., coping with changes in cognition and language, use of strategies for effective communication) and education regarding the disorder provided by relevant experts (e.g., speech-language pathologists, licensed professional counselors), separately for carepartners and individuals with progressive aphasia.

The implementation phase (Route 2, only) will allow for practice of strategies and skills learned in the first phase.

The total amount of time participants will be involved in the study will be 9 months, inclusive of follow-up.

Phase 1. Timeline for the support group portion of the study: Participants will complete pre-treatment measures during a period of 1-2 weeks prior to their first meeting. After four months of twice monthly meetings, post-treatment measures will be completed within 1-2 weeks of treatment completion. Follow-up evaluation will take place at 3-months post-treatment.

Phase 2. Timeline for the implementation/dyad training portion of the study: Post-treatment assessment from Phase 1 will serve as pre-treatment assessment for Phase 2. Treatment sessions will be held once weekly for 4 weeks, and post-treatment assessment will be completed within 1-2 weeks of phase 2 treatment completion. Follow-up evaluation will take place at 3-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

All participants must:

* speak Spanish and/or English (although participants may speak other languages in addition to Spanish and/or English)
* identify as Hispanic and/or Latinx,
* or their spouse/family member with PA identifies as Hispanic and/or Latinx
* see and hear well enough to participate
* have access to a computer or mobile device with video capability
* have an internet connection

Additional inclusion criteria for PA/ language-led dementia support group participants:

* Individuals with PA:
* Has a diagnosis of PA, or language-led dementia, and aphasia is one of the primary causes of difficulty with activities of daily living
* Aware of language difficulties and willing to discuss them
* Able to actively engage in group discussion and complete activities with minimal support
* Able to regularly attend meetings
* Willing to follow the rules of the support group for interacting with others respectfully

Additional inclusion criteria for care partner support group plus implementation phase participants:

* Individuals with PA:
* Diagnosis of aphasia or dementia that is progressive in nature, and aphasia is one of the primary causes of difficulty with activities of daily living
* Have some ability to communicate and understand communication in order to participate in training sessions
* Are functionally able to engage in training sessions (e.g., able to maintain some attention, minimal challenging behavior that would cause disruption)
* Have a care partner who also consents to participating in the project
* Care partners:
* Self-identification as a caregiver of an individual with a diagnosis of PA or language-led dementia
* Willing to discuss caregiving for individuals with PA/ language-led dementia
* Able to regularly attend meetings
* Willing to follow the rules of the support group for interacting with others respectfully

Exclusion Criteria:

• Beyond the inclusion criteria included above, no additional exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Treatment/Acceptability Survey | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  In-house Acceptability and Perception of Change Survey

SECONDARY OUTCOMES:
Acceptability Measure | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Acceptability scale for healthcare interventions (the Theoretical Framework of Acceptability based questionnaire; Sekhon et al., 2022)
% participants who complete intervention, % sessions completed | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Adherence/receipt of intervention, 0-100, greater better
% completion of homework | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Engagement, 0-100, greater better
Retention | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Number of dropouts, reasons for dropout (related to intervention or not), and overall, retention rate at final assessment and follow-up; 80% is successful at the final post-treatment assessment and 80% is successful at the 2-month follow-up, 0-100, greater better
Aphasia Impact Questionnaire | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Aphasia impact, Higher score indicates poorer quality of life (worse) Range of scores for each question: 0-4 Total 0-84
Mini-Mental State Exam | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Cognitive screener, 0-30, greater better
Quick Aphasia Battery | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Aphasia severity, 0-10, greater better
Stroke and Aphasia Quality of Life Scale- 39 | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Quality of life, greater score is better, 0-195
Progressive Aphasia Severity Scale (PASS) | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Aphasia severity, higher score = worse, 0-3
The Neuropsychiatric Inventory | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Neuropsychiatric status, higher score = worse, 0-36
Clinical Dementia Rating Scale (CDR) | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Dementia Rating, higher score = worse, 0-3
Quality of the Caregiver Patient Relationship (QCPR) | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Quality of life, higher scores is better,14-70
Dementia Quality of Life | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Quality of life, higher score is better, 28-112
Geriatric Depression Scale | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Depression, higher score is worse, 0-15
Dementia Knowledge Assessment Scale | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Dementia Knowledge, higher score is better, 0-60
Center for Epidemiologic Studies Depression Scale | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Depression, higher score is worse, 0- 60
Cuestionario de Salud 36-Item Short Form Survey Instrument | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  General health, higher score is better, 0-100
General Anxiety Disorder-7 | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Anxiety, higher score is worse, 0-21
The Duke University Religion Index | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Religion Index
Familism Scale | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Familism Scale, higher score= greater religiosity, 1-15 considering all subscales
Acculturation Rating Scale for Mexican Americans | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Acculturation, higher score is better, 20-124
Adult Carer Quality of Life Questionnaire | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Quality of Life, higher score is better, 0 -105
Brief COPE | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Coping strategies, higher score is better, 0-6
Brief Assessment Scale for Caregivers | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Coping strategies, higher score = worse, -28-28
Zarit Burden Interview | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Burden, higher score = worse, 0-88
Perceived Stress Scale | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Stress level, higher = worse, 0-40
Devereux Adult Resilience Scale | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Resilience
Dementia Management Strategies Scale (Tan et al., 2013) | Baseline, Immediately following treatment, Follow-up at 3-months post-treatment
  Dementia management, higher score= higher frequency of action, subscales 8-55

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Multilingual Lab Website — https://slhs.utexas.edu/research/multilingual-aphasia-and-dementia-research-lab/participate